CLINICAL TRIAL: NCT02827643
Title: Vitamin D and Calcium Supplement Attenuate Bone Loss Among HIV- Infected Patients Receiving Tenofovir Disoproxil Fumarate, Lamivudine or Emtricitabine and Efavirenz: An Open-label, Randomized Controlled Trial
Brief Title: Vitamin D and Calcium Supplement Attenuate Bone Loss Among HIV- Infected Patients Receiving Tenofovir Disoproxil Fumarate, Lamivudine or Emtricitabine and Efavirenz
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ID 01-59-11 ว
Record Dates: First submitted 2016-07-06; First posted 2016-07-11 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-06

CONDITIONS: Bone Density
MeSH Terms: interventions — Calcium; Ergocalciferols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TDF/3TC or FTC/EFV plus Calcium and vitamin D supplement (Active Comparator): Once daily calcium carbonate 1,250 mg that equal to elemental calcium 600 mg and weekly vitamin D2 20,000international units are given in intervention arms for duration of 24 weeks the subjects in this arm continue previous ART before enrollment to the study
  Interventions: Drug: TDF/3TC or FTC/EFV plus Calcium and vitamin D supplement
- TDF/3TC or FTC/EFV (Other): the subjects in this arm continue previous ART before enrollment to study without any intervention with standard for HIV-infected patient.
  Interventions: Other: TDF/3TC or FTC/EFV

INTERVENTIONS:
Drug: TDF/3TC or FTC/EFV plus Calcium and vitamin D supplement — Once daily calcium carbonate 1,250 mg that equal to elemental calcium 600 mg and weekly vitamin D2 20,000international units are given in intervention arms for duration of 24 weeks the subjects in this arm continue previous ART before enrollment to the study
  Other Names: ergocalciferol
  Arms: TDF/3TC or FTC/EFV plus Calcium and vitamin D supplement
Other: TDF/3TC or FTC/EFV — arm continue previous ART before enrollment to study without any intervention with standard for HIV-infected patient.
  Arms: TDF/3TC or FTC/EFV

SUMMARY:
The purpose of this study is to determine whether calcium and vitamin D supplement can attenuate bone loss in HIV-infected-patients in Thailand who receive Tenofovir disoproxil fumarate.

DETAILED DESCRIPTION:
Early initiation of antiretroviral therapy (ART) has transformed HIV infection into chronic manageable disease. Although incidence of AIDS-related mortality has decreased, it has increased for other co-morbid conditions including decrease bone mass, osteoporosis, fragility fracture. There are multi-factorial that contribute to bone loss in HIV-infected individuals including HIV virus itself that shift bone remodeling pathway toward bone resorption, lifestyle and behavioral factors, co-morbid conditions and ART.

Initiation of ART is associated with 2%-6% reduction in bone mineral density during the first 2 years of treatment regardless of ART regimens and then stabilization thereafter in the majority of the study. This magnitude of bone loss is similar to postmenopausal women during the first year.

Tenofovir disoproxil fumarate (TDF) is a nucleotide analogue reverse transcriptase inhibitor, has been associated with greater bone loss than other reverse transcriptase inhibitors, that is recommended as the first line treatment in Thailand. Nonetheless there is an evidence in western country that calcium and vitamin D supplement can attenuate bone loss in naive HIV-infected individual who start ART with TDF. Even though many experts recommend to avoid TDF and prefer abacavir, NRTIs which affect bone loss less than other NRTIs, in high fracture risk patients, more than less HIV-infected-patients can access to abacavir in resource limiting country. This research aims to study bone mineral density (BMD) in HIV infected-patient in Thai population who receive tenofovir with calcium and vitamin D supplement.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1-infected patients who start 3TC or FTC,TDF and EFV within 3 months before enrollment
* Age 18-50 years

Exclusion Criteria:

* CrCl <60mL/min/1.73 m2 ¶-
* CaCO3 supplement >500 mg/day or vitamin D supplement >800 IU/day
* Steroid used (equivalent to prednisolone> 5 mg/day more than 3 months )
* Osteoporosis treatment
* Serum Ca >10.5 g/dL
* History fragility fracture
* Pregnancy or breastfeeding
* Secondary amenorrhea
* Hyperthyroidism
* History of kidney stone
* Current active opportunistic infection

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-03 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
percentage change of bone density | 24 weeks

SECONDARY OUTCOMES:
change in 25(OH)D level | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Patawee Boontanondha, Faculty of Medicine Ramathibodi Hospital, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes